CLINICAL TRIAL: NCT05703555
Title: INTRUSION: Unraveling the INTRatUmoral PK/PD relatION for SAR408701
Acronym: INTRUSION
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the decision to discontinue the global clinical development program of tusamitamab ravtansine
Sponsor: Erasmus Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Debbie Robbrecht, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INTRUSION; 2022-003451-34 (EudraCT Number)
Record Dates: First submitted 2022-12-13; First posted 2023-01-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Lung Cancer; Metastatic Breast Cancer; Metastatic Gastric Cancer
Keywords: tusamitamab ravtansine; CEACAM5; Pharmacokinetics
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Stomach Neoplasms | interventions — tusamitamab ravtansine

STUDY DESIGN:
Intervention Model Description: open-label, multi-cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tusamitamab ravtansine 100mg/m2 (Experimental): Tusamitamab ravtansine 100 mg/m2 IV Q2W
  Interventions: Drug: Tusamitamab ravtansine

INTERVENTIONS:
Drug: Tusamitamab ravtansine — Eligible subjects will receive Tusamitamab ravtansine (100mg/m2 IV Q2W). Subjects without evidence of disease progression or drug related toxicity can continue treatment with Tusamitamab ravtansine (100 mg/m2 IV Q2W) until disease progression, unacceptable toxicity occurs, or the participant's or Investigator's decision to stop the treatment.
  Other Names: SAR408701

SUMMARY:
This study is a prospective, open-label, multi-cohort, exploratory phase II clinical trial in patients with either CEACAM5-positive NSQ NSCLC, ER+ breast cancer or gastric cancer. Eligible subjects will receive Tusamitamab ravtansine (100mg/m2 IV Q2W). The investigators hypothesize that intratumoral exposure of Tusamitamab ravtansine would be an important factor in determining treatment efficacy. Combining exposure with measurements of tumor PD reactions in a proper PK/PD study is the goal of this study.

DETAILED DESCRIPTION:
The investigators hypothesize that intratumoral exposure of Tusamitamab ravtansine would be an important factor in determining treatment efficacy. The rationale to develop an antibody-drug conjugate, like tusamitamab ravtansine, is that it concentrates the active compound (DM4) in cancer tissues, thus confirming this hypothesis in human subjects would be an important step forward. Combining exposure with measurements of tumor PD reactions in a proper PK/PD study is the goal of the study.

Tusamitamab ravtansine is being developed in NSQ NSCLC. The results of the first-in-human study in NSQ NSCLC patients were promising and participants could thus benefit from this treatment. However, other tumor types also express CEACAM5 in tumor cells. The investigators will also recruit metastatic ER+ breast cancer patients and metastatic gastric cancer patients. Hence, there has been more limited data on the safety and efficacy in this patient populations. Addition of these cohorts will help to understand the influence of primary tumor type in determining intratumoral concentrations of Tusamitamab ravtansine.

CEACAM5-positive is defined as IHC ≥2+ in intensity in ≥50% of the tumor cells expressing CEACAM5. Yet, the cut-off value for CEACAM5 expression is arbitrarily selected. A PK/PD relation between CEACAM5 expression and exposure would support the current applied cut-off value for CEACAM5 expression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18y) at the time of signing the Informed Consent Form (ICF).
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Estimated life expectancy ≥ 3 months
* Expression of CEACAM5 established by an IHC assay of ≥2+ in intensity involving at least 50% of the tumor cell population in archival tumor sample (or, if not available, a fresh biopsy sample) at a metastatic site (mandatory) including distant lymph nodes.
* Either: Metastatic or irresectable Non-Squamous Non-Small Cell Lung Cancer without EGFR/ALK/ROS aberration, as diagnosed by histological evaluation, after chemotherapy (restricted to 1 line of platinum-based chemotherapy) and immunotherapy (not more than 1 line). These therapies may have been applied concurrent or sequential; Or: Metastatic ER+ breast cancer, pathologically confirmed. ER+ is defined as ≥1% tumor staining by IHC. Participants must be no longer eligible for hormonal therapy. Participants may have had at maximum 1 prior systemic chemotherapy line.

A chemotherapy line in advanced/metastatic disease is an anti-cancer regimen that contains at least 1 cytotoxic chemotherapy agent and was discontinued due to progression. If a cytotoxic chemotherapy regimen was discontinued for a reason other than disease progression then this regimen does not count as a "prior line of chemotherapy" unless this regimen was discontinued after at least 2 cycles of treatment.

Or: Metastatic gastric cancer, pathologically confirmed, with no regular treatment options left and having received all standard of care treatments.

* Metastatic lesion accessible for repeated biopsy and willingness to undergo sequential biopsies.
* Lesion to be biopsied must be measurable on CT according to RECIST v1.1.
* Ability and willingness to give written informed consent and to comply with the requirements of the study.

Exclusion Criteria:

Medical conditions:

* History within the last 3 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* Symptomatic or untreated brain metastases or history of leptomeningeal disease. Participants with previously treated brain metastases may participate provided that:

  i. metastases are stable for at least 4 weeks according to imaging and symptoms returned to baseline; ii. there is no evidence of new or enlarging brain metastases; iii. the participant does not require any corticosteroids to manage brain metastases within 3 weeks prior to the first dose of study intervention.
* Recent (within 6 months) Pulmonary Embolism or other recent (within 6 months) thromboembolic event requiring anticoagulant therapy.
* Ascites requiring palliative intervention such as repeated drainage.
* Prior toxicity incurred as a result of previous anti-cancer therapy (radiation therapy, chemotherapy, or surgery) that have not resolved to ≤ grade 2 according to NCI-CTCAE version 5.0 [Appendix 3] except ocular toxicity, this should be grade 0 at baseline, without the exception of alopecia, vitiligo, or active thyroiditis controlled with hormone replacement therapy.
* Major surgical procedure (including open biopsy and excluding central line intravenous catheter) within 28 days prior to Cycle 1 Day 1, or anticipation of the need for major surgery during the course of the study treatment.
* History of human immunodeficiency virus (HIV) antibody positive or use of antiretroviral therapy. No HIV testing is required unless mandated by local health authority.
* Medical conditions requiring concomitant administration of strong CYP3A inhibitor or inducer unless it can be discontinued at least 2 weeks before the first administration of study intervention and discontinued for the duration of the study intervention.
* Unable or unwilling to stop the use of (herbal) supplements which can strongly induce or inhibit CYP3A, including grapefruit containing food or juice or St. John's Wort from 2 weeks before the first Tusamitamab ravtansine administration up to the last Tusamitamab ravtansine administration.
* Medical condition requiring concomitant administration of medication with a narrow therapeutic window that is metabolized by cytochrome P450 (CYP450) from 2 weeks before the first Tusamitamab ravtansine administration up to the last Tusamitamab ravtansine administration. See also section 5.2.

Specific Tusamitamab ravtansine (SAR408701) related conditions:

* Less than 4 weeks or less than 5 times the half-life, whichever is shorter, since the last treatment of chemotherapy, biological therapy, immunotherapy or systemic radiotherapy (except palliative radiation delivered to <20% of bone marrow), before Cycle 1 Day 1.
* Current or recent (within 4 weeks prior to Cycle 1 Day 1) treatment with another Investigational Product or participation in another investigational interventional study.
* Any prior therapy targeting CEACAM5.
* Prior maytansinoid DM4 treatment (ADC).
* Unresolved corneal disorder or any previous corneal disorder considered by an ophthalmologist to predict higher risk of drug-induced keratopathy.
* Use of contact lenses: Participants using contact lenses who are not willing to stop wearing them for the duration of the study intervention are excluded.
* Unresolved grade ≥0 ocular symptoms according to NCI-CTCAE version 5.0 [Appendix 3].
* Unresolved grade ≥2 motor or sensory neuropathy symptoms according to NCI-CTCAE version 5.0 [Appendix 3].
* Known hypersensitivity to any of the Investigational Product's excipients.
* Concurrent treatment with any other anti-cancer therapy.
* Previous enrollment in this study or current participation in any other clinical study involving an investigational study treatment or any other type of medical research.

Diagnostic assessments:

* Inadequate bone marrow function, as defined by any of the following:

  * Absolute Neutrophil Count (ANC) < 1.5 x 109/L.
  * Platelet count < 100 x 109/L.
  * Hemoglobin < 6.0 mmol/L (<9.6 g/dL).
  * No blood and blood product transfusion or growth factors within two weeks prior to Cycle 1 Day 1.
* Inadequate liver function, as defined by any of the following:

  * Serum (total) bilirubin > 1.5 x the Upper Limit of Normal (ULN) for the institution if no liver metastases (> 2 x ULN in patients with liver metastases).
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase (AP) > 2.5 x ULN if no liver metastases (> 5x ULN in participants with liver metastases and for participants with bone metastases AP ≤ 5 ULN is allowed).
  * Hepatitis B surface antigen or hepatitis C positivity in combination with abnormal liver function tests if it is indicated to be determined by the Investigator.
* Inadequate renal function, as defined by any of the following:

  * Serum creatinine > 1.5 x ULN.
  * Estimated Glomerular Filtration Rate of < 50 mL/min/1.73m2 as estimated using CKD-EPI formula.
* Serum albumin value < 25 g/L

Others:

* Patients who are pregnant or breastfeeding. Female participants of childbearing potential must have a negative serum pregnancy test before the first dose of study intervention. Serum pregnancy tests will be carried out every 4 weeks during study treatment.
* Absence of effective means of contraception on Cycle 1 Day 1 in female participants of childbearing potential (defined as <2 years after last menstruation and not surgically sterile).
* Male participants who are not surgically sterile and for least 4 months after the last dose of study intervention:

I. do not agree to be abstinent for sexual intercourse; or II. do not agree to use a male condom when engaging in sexual activity that allows for passage of ejaculate to another person; or III. donate sperm and do not refrain from donating sperm.

* Individuals accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalized.
* History of drug or alcohol abuse in the opinion of the Investigator within 3 years before screening.
* Evidence of any other medical condition (such as psychiatric illness, infectious diseases, physical examination or laboratory findings) that may interfere with the planned treatment, affect patient compliance or place the patient at high risk for treatment-related complications, as judged by the Investigator.
* Patients on anticoagulants for whom temporarily stop and start is not an option to obtain biopsies, at the discretion of the investigator and/or per local standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
intratumoral DM4 concentration | approximately 5 weeks, more specific day 3 of cycle 2 (each cycle is 14 days)
  Intratumoral DM4 exposure, as measured in a biopsied lesion using a PK assay.

SECONDARY OUTCOMES:
Intratumoral tusamitamab ravtansine concentration | approximately 5 weeks, more specific day 3 of cycle 2 (each cycle is 14 days)
  Intratumoral concentrations of Tusamitamab ravtansine and metabolites of DM4: Lys-SPDB-DM4, Me-DM4 using a PK assay
Incidence of grade 3 or 4 adverse events | during treatment (up to 2 years and 12 weeks)
  Incidence of grade 3 or 4 adverse events as assessed by CTCAE version 5.0
Response to treatment | every 8 weeks during treatment (up to 2 years and 12 weeks)
  Number of participants with either progressive disease, stable disease, partial response or complete response according to RECIST v 1.1
CEACAM5 expression | approximately 5 weeks, more specific day 3 of cycle 2 (each cycle is 14 days)
  Change in CEACAM5 expression from baseline as assessed by immunohistochemistry
RNA expression levels | approximately 5 weeks, more specific day 3 of cycle 2 (each cycle is 14 days)
  Change from baseline in RNA expression levels as assessed with differential gene-level analysis in DESeq2
circulating CEA levels | every 8 weeks during treatment (up to 2 years and 12 weeks)
  Number of patients with elevated levels of circulation CEA
tumor genomic features | baseline
  Somatic copy number, strucural and nucleotide alterations as assessed by whole genome sequencing
Maximal plasma concentration | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  Cmax and its corresponding time (Tmax)
AUCinf | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  AUCinf - Area under the curve form time of dosing extrapolated to infinity of AUC0-t + Clast/lambda z
AUClast | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  AUClast - Area under the curve form the time of dosing to the time of the last quantifiable concentration calculated using the linear trapezoidal rule
AUCt | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  AUCt - Area under the concentration versus time curve
Thalf | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  Thalf will be calculated as ln(2)/Lambda z
systemic tusamitamab ravtansine concentration | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  Clearance (Cl)
Volume of distribution | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  Volume of distribution
concentration DM4 metabolites: Lys-SPDB-DM4, Me-Dm4 | baseline and at 7 different time points during treatment (3x cycle 1 day 1, 1x pre-dose cycle 2 day 1, 2x cycle 2 day 2, and 1x pre-dose cycle 4 day 1) (each cycle is 14 days)
  concentration of metabolites of DM4 will be described
features in tumor micro-environment | approximately 5 weeks, more specific day 3 of cycle 2 (each cycle is 14 days)
  RNA-sequencing to deduce the immune contexture using quanTIseq, tumor infiltrating lymphocyte signatures and related workflows

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Robbrecht, Dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
By means of a publication in a peer-reviewed international journal
Supporting Information: Study Protocol
Time Frame: Within 12 months of last visit of last patient